CLINICAL TRIAL: NCT02110888
Title: Subcutaneous Peripheral Nerve Stimulation (PNS) as "Hybrid Stimulation" After Failure of Spinal Cord Stimulation (SCS) to Control the Back Pain Component in Failed Back Surgery Syndrome (FBSS) Patients.(CUMPNS Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUMPNS
Record Dates: First submitted 2014-04-04; First posted 2014-04-10 (Estimated); Last update posted 2021-10-18 (Actual); Status verified 2021-09

CONDITIONS: Failed Back Surgery Syndrome
MeSH Terms: conditions — Failed Back Surgery Syndrome

ARMS (2):
- SCS + PNS (Experimental): Mutlticolumn SCS lead + Monocolumn SCS lead
  Interventions: Device: Subcutaneous peripheral nerve stimulation
- SCS (Active Comparator): Mutlticolumn SCS lead
  Interventions: Other: SCS Only

INTERVENTIONS:
Device: Subcutaneous peripheral nerve stimulation
  Arms: SCS + PNS
Other: SCS Only
  Arms: SCS

SUMMARY:
Despite globally favourable outcomes of Spinal Cord Stimulation (SCS), a significant proportion of Failed Back Surgery Syndrome (FBSS) patients do not obtain adequate coverage of low back pain. Peripheral Nerve Stimulation (PNS) has obtained the European Conformity mark for the treatment of chronic refractory neuropathic pain and is now commonly used in some countries to target back pain. However, the potential value of combining SCS and PNS as "hybrid stimulation" remains poorly described with only isolated case reports or limited experience in various indications.

The "CUMPNS" comparative randomized study is designed to demonstrate the potential analgesic efficacy of PNS in addition to previously implanted SCS, to treat the residual low back pain component pain in refractory FBSS patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 80 years.
* History of FBSS after one or more surgical procedures on the spine, treated with SCS,
* Failure of well conducted conservative treatment (drug or non-drug).
* Patients implanted with a single-column or multicolumn SCS lead providing significant relief of the radicular pain component.
* Persistent failure on the low back pain component despite the efficacy of SCS on the radicular pain component.
* Patients with documented residual neuropathic low back pain (DN4, sensorimotor studies, clinical examination, pain characteristics, etc.).
* Patients with significant residual low back pain with mean intensity on Visual Analogue Scale (VAS) ≥ 40 mm) despite Conventional Medical Management (CMM) and SCS (mean measure calculated on daily VAS scores on 5 consecutive days).
* Positive response to Transcutaneous Electrical Nerve Stimulation (TENS) trial on the back pain component.
* Patients understanding and accepting the study constraints.
* Patients covered by French national health insurance.
* Patients have signed the Informed Consent Form after being provided with clear and honest information about the study.
* Absence of active psychosis or serious psychotic history requiring hospitalisation.
* Absence of active cancer.

Exclusion Criteria:

* Age < 18 years and > 80 years.
* Back pain amenable to further aetiological biomechanical surgery (discogenic pain, spinal instability, spinal deformity, etc.).
* Surgical, psychiatric or anaesthetic contraindication to PNS lead implantation.
* Negative response to TENS trial.
* Absence of signature of the informed consent form.
* Patients not covered by French national health insurance.
* Subjects requiring closer protection, i.e. minors, pregnant women, nursing mothers, subjects deprived of their freedom by a court or administrative decision, subjects admitted to a health or social welfare establishment, major subjects under legal protection, and finally patients member of a high-risk population.
* Women of childbearing age not using effective contraception.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2018-10-14 (Actual); Study Completion 2018-10-14 (Actual)

PRIMARY OUTCOMES:
Relative change of low back pain surface (expressed as a percentage, %) | 3 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Philippe RIGOARD, MD, PhD, Principal Investigator — Poitiers University Hospital
Locations (1):
- Poitiers University Hospital, Poitiers, France